CLINICAL TRIAL: NCT01280903
Title: Promoting Physical Activity in Older Adults With Comorbidity
Brief Title: Staying Active With Arthritis: RCT of Physical Activity for Older Adults With Osteoarthritis and Hypertension
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Elizabeth Schlenk, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO09110029; R01NR010904-01A1 (NIH)
Record Dates: First submitted 2010-12-17; First posted 2011-01-21 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee; Hypertension
Keywords: Osteoarthritis, Knee; Hypertension; Exercise; Physical activity; Self Efficacy; Patient Compliance; Aged
MeSH Terms: conditions — Osteoarthritis, Knee; Hypertension; Motor Activity; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STAR Intervention (Experimental): Staying Active with Arthritis Intervention
  Interventions: Behavioral: STAR Intervention
- Attention-Control (Placebo Comparator): Senior Health Information Intervention
  Interventions: Behavioral: Attention-Control

INTERVENTIONS:
Behavioral: STAR Intervention — The 24-week modified Staying Active with Arthritis (STAR) intervention, guided by self-efficacy theory and modified to address comorbid hypertension, consists of 6 weekly individual face-to-face exercise sessions by a licensed physical therapist, 9 biweekly telephone counseling sessions by a registered nurse to continue the use of self-efficacy strategies, and lower extremity exercise and fitness walking being carried out at home between sessions. There will be no contact with participants during weeks 7, 9, 11, 13, 15, 17, 19, 21, and 23. During the 6-month follow-up period, the participants will be contacted briefly by telephone by a registered nurse at weeks 30, 36, and 48 for a general check-up.
  Arms: STAR Intervention
Behavioral: Attention-Control — Attention-Control is a 24-week general health education program for older adults that consists of 6 weekly telephone sessions by a registered nurse followed by 9 biweekly telephone sessions by a registered nurse. There will be no contact with participants during weeks 7, 9, 11, 13, 15, 17, 19, 21, and 23. Topics include cancer screenings; immunizations; osteoporosis; low vision; hearing loss; talking with your primary care provider; eating healthy (two parts); sleep and aging; injury prevention (two parts: balance problems and falls); oral health; foot care; and mental health (depression). During the 6-month follow-up period, the participants will be contacted briefly by telephone by a registered nurse at weeks 30, 36, and 48 for a general check-up.
  Arms: Attention-Control

SUMMARY:
The purpose of the Staying Active with Arthritis (STAR) research study is to determine if a 6-month program will improve leg exercise, fitness walking, and clinical outcomes (function, blood pressure, leg strength, pain, fatigue, and health-related quality of life) in older adults with osteoarthritis of the knee and high blood pressure.

DETAILED DESCRIPTION:
Over 9 million Americans have symptomatic osteoarthritis (OA) of the knee, a chronic disease associated with frequent joint pain, functional limitations, and quadriceps weakness that intrude upon everyday life. At least half of those with OA of the knee are diagnosed with hypertension or high blood pressure (HBP), one of the most prevalent risk factors for cardiovascular disease. Many other individuals with OA of the knee unknowingly have HBP and remain untreated. Our own work and that of others suggest that persons with OA of the knee experience reductions in BP when they participate in a regular regimen of physical activity. Even small decreases in systolic and diastolic BP found with physical activity are clinically significant, e.g., a 2 mm Hg decrease reduces the risk of stroke by 14% - 17%, and the risk of coronary heart disease is reduced by 6% - 9%. Yet, only 15% of persons with OA and 47% with HBP engage in regular physical activity. The purpose of this study is to investigate how the individually delivered, home-based, 6-month modified Staying Active with Arthritis (STAR) intervention, guided by self-efficacy theory and modified to address comorbid HBP, affects lower extremity exercise (flexibility, strengthening, and balance), fitness walking, functional status, BP, quadriceps strength, pain, fatigue, and health-related quality of life (HRQoL) in a convenience sample of 224 adults age 50 years or older with OA of the knee and HBP. Using a randomized controlled, 2-group design, we (1) hypothesize that at the end of the 6-month intervention period and 6 months after the intervention period ends those who receive the modified STAR intervention will be more likely to perform lower extremity exercise, participate in fitness walking, show improvements in objective functional status, and demonstrate reductions in BP than those who receive attention-control. Secondarily, we will (2) evaluate the impact of the modified STAR intervention, compared to attention-control, on subjective functional status, quadriceps strength, pain, fatigue, and HRQoL at both time points; (3) explore the impact of the modified STAR intervention, compared to attention-control, on self-efficacy and outcome expectancy at both time points; (4) explore the relationship between self-efficacy and outcome expectancy; and (5) explore the extent to which self-efficacy and outcome expectancy mediate the relationship between the modified STAR intervention and performance of lower extremity exercise and participation in fitness walking. Data will be analyzed using repeated measures modeling.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older.
* Is community dwelling.
* Has osteoarthritis of the knee.
* Has hypertension for which monotherapy or combination pharmacological treatment is prescribed.
* Able to complete a behavioral run-in consisting of completing questionnaires, using a 7-day electronic-diary, and wearing an ActiGraph accelerometer at the waist for 7 days.
* Has written permission to participate from the physician.

Exclusion Criteria:

* Reports currently doing lower extremity exercise => 2 times/week.
* Reports currently fitness walking => 90 minutes/week.
* Incapable of managing their own treatment regimen.
* Does not have, or cannot use, a telephone or is unwilling to provide a telephone number.
* Has received cortisone or Synvisc injections in the knee, angioplasty, stents, or a pacemaker in the past 6 months.
* Reports unstable cardiovascular, pulmonary, or metabolic disease or signs and symptoms suggestive of cardiovascular, pulmonary, or metabolic disease that restrict activity.
* Has resting systolic blood pressure => 160 mm Hg or diastolic blood pressure => 100 mm Hg.
* Reports other conditions, such as osteoarthritis of the hip, spinal stenosis, inflammatory arthritis, foot drop, diabetes treated with insulin, or diabetic complications that may affect performance of lower extremity exercise and participation in fitness walking.
* Reports current knee conditions, such as meniscus tears and knee ligament ruptures.
* Reports major depression that may impact the ability to fully participate in this study.
* Is scheduled to undergo a major surgical procedure in the next 13 months.
* Is concurrently participating in a drug or psychoeducational trial that may confound, or be confounded by, participation in this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Schlenk, PhD, RN, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Nursing, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schlenk EA, Sereika SM, Martire LM, Shi X. Older adults' social network and support and its association with physical activity. Geriatr Nurs. 2021 Mar-Apr;42(2):517-523. doi: 10.1016/j.gerinurse.2020.09.006. Epub 2020 Oct 7. PMID 33039202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | STAR Intervention | Attention-Control
Started | 91 | 91
Completed | 68 (91 participants analyzed per intention-to-treat) | 75 (91 participants analyzed per intention-to-treat)
Not Completed | 23 | 16
Not completed — Lost to Follow-up | 23 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STAR Intervention | Attention-Control | Total
Number analyzed (Participants) | 91 | 91 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.47 (8.46) | 64.96 (7.76) | 64.71 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 66 | 133
  Male | 24 | 25 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 88 | 88 | 176
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 15 | 32
  White | 66 | 66 | 132
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 91 | 91 | 182
Body mass index [Mean (Standard Deviation); unit: kg/m²] | 34.50 (7.48) | 33.64 (6.43) | 34.07 (6.97)
Number of comorbidities [Mean (Standard Deviation); unit: comorbidities] | 6.8 (2.9) | 6.5 (2.7) | 6.6 (2.8)
Marital status [Number; unit: participants]
  Married | 38 | 46 | 84
  Not married | 53 | 45 | 98
Educational status [Number; unit: participants]
  > High school | 72 | 71 | 143
  High school or less | 19 | 19 | 39
  Missing | 0 | 1 | 0
Employment status [Number; unit: participants]
  Employed | 45 | 43 | 88
  Not employed | 46 | 48 | 94
Household income [Number; unit: participants]
  < $50,000/year | 37 | 38 | 75
  $50,000 or more/year | 39 | 38 | 77
  Missing | 15 | 15 | 30
Lower extremity exercise (e-diary): days/week [Mean (Standard Deviation); unit: days/week] | 0.41 (1.01) | 0.36 (1.02) | 0.38 (1.01)
Lower extremity exercise (e-diary): minutes/week [Mean (Standard Deviation); unit: minutes/week] | 7.60 (24.87) | 7.43 (24.51) | 7.52 (24.52)
Lower extremity exercise (e-diary): average minutes/day [Mean (Standard Deviation); unit: average minutes/day] | 1.09 (3.55) | 1.06 (3.47) | 1.07 (3.50)
Lower extremity exercise (e-diary): volume [repetitions x sets over 7-day period]/week [Mean (Standard Deviation); unit: repetitions x sets/week] | 56.93 (255.39) | 30.41 (121.21) | 43.67 (199.79)
Fitness walking (e-dairy): days/week [Mean (Standard Deviation); unit: days/week] | 0.65 (1.41) | 0.57 (1.31) | 0.61 (1.36)
Fitness walking (e-diary): minutes/week [Mean (Standard Deviation); unit: minutes/week] | 18.54 (47.45) | 15.33 (37.83) | 16.93 (42.82)
Fitness walking (e-diary): average minutes/day [Mean (Standard Deviation); unit: average minutes/day] | 2.65 (6.78) | 2.19 (5.40) | 2.42 (6.12)
Activity minutes over 7 days (ActiGraph): no to very low (counts of 0-99/min) [Mean (Standard Deviation); unit: minutes] | 3155.5 (714.6) | 2934.8 (842.3) | 3045.2 (786.7)
Activity minutes over 7 days (ActiGraph): light (counts of 100-2,019/min) [Mean (Standard Deviation); unit: minutes] | 2348.7 (572.0) | 2418.8 (632.1) | 2383.8 (602.2)
Activity minutes over 7 days (ActiGraph): moderate-to-vigorous (counts of > 2,020/min) [Mean (Standard Deviation); unit: minutes] | 275.8 (154.0) | 365.5 (288.4) | 320.6 (234.9)
Number of bouts over 7 days (ActiGraph): bouts of moderate-to-vigorous activity [Mean (Standard Deviation); unit: bouts] | 1.7 (2.6) | 2.7 (6.5) | 2.2 (5.0)
Mean duration of bouts over 7 days (ActiGraph): bouts of moderate-to-vigorous activity n=96 [Mean (Standard Deviation); unit: minutes] — Population: Some participants in each group had no bouts at baseline of => 10 consecutive minutes participating in activity at the => 2,020 counts threshold.
  minutes
    number analyzed (Participants) | 45 | 51 | 96
    (all) | 17.2 (7.5) | 19.9 (8.7) | 18.6 (8.2)
Mean number of daily activity minutes (ActiGraph): no to very low (counts of 0-99/min) [Mean (Standard Deviation); unit: minutes] | 440.14 (96.5) | 410.26 (111.1) | 425.2 (104.9)
Mean number of daily activity minutes (ActiGraph): light (counts of 100-2,019/min) [Mean (Standard Deviation); unit: minutes] | 327.5 (76.8) | 339.3 (86.4) | 333.4 (81.7)
Mean number of daily activity minutes (ActiGraph): moderate-to-vigorous (counts of >2,020/min) [Mean (Standard Deviation); unit: minutes] | 38.3 (20.7) | 51.2 (38.7) | 44.7 (31.6)
Mean number of daily bouts (ActiGraph): bouts of moderate-to-vigorous activity [Mean (Standard Deviation); unit: bouts] | 0.2 (0.4) | 0.4 (0.9) | 0.3 (0.7)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 122.09 (15.01) | 121.82 (13.78) | 121.96 (14.37)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 72.86 (11.18) | 73.15 (9.47) | 73.01 (10.33)
6-minute walk [Mean (Standard Deviation); unit: yards] | 486.2 (105.9) | 484.7 (88.1) | 485.5 (97.1)
Short Physical Performance Battery: total [Mean (Standard Deviation); unit: units on a scale] — Subscale scores are summed for a total scale score; the total scale score range is 0-13; higher scores are better
  units on a scale | 11.0 (1.7) | 10.6 (1.6) | 10.8 (1.6)
Short Physical Performance Battery: repeated chair stands [Mean (Standard Deviation); unit: units on a scale] — The repeated chair stands subscale score range is 0-4; higher scores are better
  units on a scale | 2.9 (1.2) | 2.7 (1.1) | 2.8 (1.1)
Short Physical Performance Battery: 4-meter usual walk [Mean (Standard Deviation); unit: units on a scale] — The 4-meter usual walk subscale score range is 0-4; higher scores are better
  units on a scale | 4.0 (0.2) | 4.0 (0.0) | 4.0 (0.2)
Short Physical Performance Battery: standing balance [Mean (Standard Deviation); unit: units on a scale] — The standing balance subscale score range is 0-5; higher scores are better
  units on a scale | 4.2 (0.8) | 4.0 (0.9) | 4.1 (0.8)
Chair sit-and-reach [Mean (Standard Deviation); unit: inches] | -1.4 (5.7) | -0.8 (5.6) | -1.1 (5.6)
8-foot up-and-go [Mean (Standard Deviation); unit: seconds] | 6.5 (1.8) | 6.6 (1.3) | 6.6 (1.6)
Quadriceps strength (mean maximum for right and left quadriceps) [Mean (Standard Deviation); unit: pounds] | 41.8 (13.5) | 43.0 (16.1) | 42.4 (14.8)
Western Ontario and McMaster Universities Osteoarthritis Index: Pain [Mean (Standard Deviation); unit: units on a scale] — The WOMAC Osteoarthritis Index Pain subscale score range is 0-20; lower scores are better
  units on a scale | 5.8 (3.9) | 4.8 (3.0) | 5.3 (3.5)
Western Ontario and McMaster Universities Osteoarthritis Index: Function [Mean (Standard Deviation); unit: units on a scale] — The WOMAC Osteoarthritis Index Function subscale score range is 0-68; lower scores are better
  units on a scale | 22.5 (13.4) | 19.3 (11.9) | 20.9 (12.8)
Western Ontario and McMaster Universities Osteoarthritis Index: Stiffness [Mean (Standard Deviation); unit: units on a scale] — The WOMAC Osteoarthritis Index Stiffness subscale score range is 0-8; lower scores are better
  units on a scale | 3.1 (1.8) | 2.7 (1.8) | 2.9 (1.8)
Short Form-36v2 Health Survey: Bodily Pain [Mean (Standard Deviation); unit: units on a scale] — The subscale score range is 0-100; higher scores are better
  units on a scale | 55.7 (20.3) | 56.8 (18.7) | 56.2 (19.5)
Short Form-36v2 Health Survey: Physical Functioning [Mean (Standard Deviation); unit: units on a scale] — The subscale score range is 0-100; higher scores are better
  units on a scale | 62.0 (23.4) | 65.2 (19.7) | 63.6 (21.6)
Short Form-36v2 Health Survey: Physical Component Score [Mean (Standard Deviation); unit: units on a scale] — This summary scale is composed of eight subscale scores primarily derived from the physical functioning, role functioning-physical, and bodily pain scores; the scale score range is 0-100; higher scores are better
  units on a scale | 42.0 (8.8) | 42.8 (8.6) | 42.4 (8.7)
Short Form-36v2 Health Survey: Mental Component Score [Mean (Standard Deviation); unit: units on a scale] — This summary scale is composed of eight subscale scores primarily derived from the mental health, role functioning-emotional, and social functioning scores; the scale score range is 0-100; higher scores are better
  units on a scale | 53.4 (9.8) | 54.0 (9.4) | 53.7 (9.6)
Brief Fatigue Inventory [Mean (Standard Deviation); unit: units on a scale] — The scale score range is 0-10; lower scores are better
  units on a scale | 2.8 (2.6) | 2.7 (2.2) | 2.8 (2.4)
Self-efficacy: Exercise [Mean (Standard Deviation); unit: units on a scale] — The subscale score range is 0-100; higher scores are better
  units on a scale | 72.8 (28.0) | 74.4 (27.2) | 73.6 (27.5)
Self-efficacy: Exercise Barriers [Mean (Standard Deviation); unit: units on a scale] — The subscale score range is 0-100; higher scores are better
  units on a scale | 60.3 (25.6) | 68.3 (21.4) | 64.3 (23.9)
Self-efficacy: Arthritis Pain [Mean (Standard Deviation); unit: units on a scale] — The subscale score range is 10-100; higher scores are better
  units on a scale | 73.7 (17.0) | 74.4 (18.2) | 74.1 (17.6)
Self-efficacy: Arthritis Function [Mean (Standard Deviation); unit: units on a scale] — The subscale score range is 10-100; higher scores are better
  units on a scale | 83.1 (15.5) | 85.2 (15.6) | 84.2 (15.6)
Self-efficacy: Arthritis Other Symptoms [Mean (Standard Deviation); unit: units on a scale] — The subscale score range is 10-100; higher scores are better
  units on a scale | 76.8 (17.4) | 77.8 (17.2) | 77.3 (17.2)
Perceived Therapeutic Efficacy - Exercise & Arthritis [Mean (Standard Deviation); unit: units on a scale] — The PTE Exercise & Arthritis scale score range is 0-100; higher scores are better
  units on a scale | 67.8 (24.5) | 72.1 (21.7) | 70.0 (23.1)
Perceived Therapeutic Efficacy - Exercise & Hypertension [Mean (Standard Deviation); unit: units on a scale] — The PTE Exercise & Hypertension scale score range is 0-100; higher scores are better
  units on a scale | 74.2 (21.2) | 74.7 (23.4) | 74.5 (22.3)

OUTCOME MEASURES:

1. Primary Outcome: Performance of Lower Extremity Exercise at 25 Weeks
Description: Measured by the electronic-diary in terms of the total volume of lower extremity exercise (i.e., the number of days the participant reports completing a lower extremity exercise session and the total number of lower extremity exercises per day performed [repetitions x sets] over a 7-day period).
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: repetitions x sets/week
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
repetitions x sets/week | 46.84 (4.59) | 1.90 (0.86)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p < .0001, Mixed Models Analysis

2. Primary Outcome: Participation in Fitness Walking at 25 Weeks
Description: Measured by the ActiGraph accelerometer in terms of mean daily activity minutes of none to very low, light, and moderate-to-vigorous activity counts summarized over a 7-day period.
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: minutes
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
minutes
  None to very low | 434.89 (11.69) | 409.98 (11.54)
  Light | 314.07 (9.29) | 321.44 (9.18)
  Moderate-to-vigorous | 40.53 (2.68) | 46.69 (3.93)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.130, Mixed Models Analysis — p=0.130 for None to very low
Statistical Analysis 2: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.573, Mixed Models Analysis — p=0.573 for Light
Statistical Analysis 3: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.197, Mixed Models Analysis — p=0.197 for Moderate-to-vigorous

3. Primary Outcome: Objective Functional Status by the 6-minute Walk at 25 Weeks
Description: Measured by the 6-minute walk (yards) as part of the performance-based functional status assessment.
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: yards
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
yards | 465.46 (18.82) | 483.02 (14.47)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.461, Mixed Models Analysis

4. Primary Outcome: Objective Functional Status by the Short Physical Performance Battery at 25 Weeks
Description: Measured by the Short Physical Performance Battery (total scale score) as part of the performance-based functional status assessment; subscale scores are summed for a total scale score; the scale score range is 0-13; higher scores are better.
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale | 11.29 (0.22) | 10.86 (0.23)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.180, Mixed Models Analysis

5. Primary Outcome: Systolic Blood Pressure at 25 Weeks
Description: Measured by the OMRON HEM-907XL automatic professional digital blood pressure monitor in mm Hg.
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
mm Hg | 120.33 (1.74) | 123.07 (1.68)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.258, Mixed Models Analysis

6. Primary Outcome: Diastolic Blood Pressure at 25 Weeks
Description: Measured by the OMRON HEM-907XL automatic professional digital blood pressure monitor in mm Hg.
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
mm Hg | 71.74 (1.20) | 73.10 (1.16)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.416, Mixed Models Analysis

7. Primary Outcome: Performance of Lower Extremity Exercise at 52 Weeks
Description: Measured by the electronic-diary in terms of the total volume of lower extremity exercise (i.e., the number of days the subject reports completing a lower extremity exercise session and the total number of lower extremity exercises per day performed [repetitions x sets] over a 7-day period).
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: repetitions x sets/week
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
repetitions x sets/week | 42.06 (6.74) | 3.14 (1.22)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p < .0001, Mixed Models Analysis

8. Primary Outcome: Participation in Fitness Walking at 52 Weeks
Description: as for outcome 2
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: minutes
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
minutes
  None to very low | 426.71 (11.97) | 408.30 (11.70)
  Light | 318.04 (9.50) | 321.01 (9.30)
  Moderate-to-vigorous | 39.37 (2.74) | 47.97 (3.97)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.272, Mixed Models Analysis — p=0.272 for None to very low
Statistical Analysis 2: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.823, Mixed Models Analysis — p=0.823 for Light
Statistical Analysis 3: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.076, Mixed Models Analysis — p=0.076 for Moderate-to-vigorous

9. Primary Outcome: Objective Functional Status by the 6-minute Walk at 52 Weeks
Description: Measured by the 6-minute walk (yards) as part of the performance-based functional status assessment.
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: yards
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
yards | 480.29 (16.89) | 465.36 (19.26)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.561, Mixed Models Analysis

10. Primary Outcome: Objective Functional Status by the Short Physical Performance Battery at 52 Weeks
Description: as for outcome 4
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale | 11.20 (0.24) | 11.25 (0.19)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.856, Mixed Models Analysis

11. Primary Outcome: Systolic Blood Pressure at 52 Weeks
Description: Measured by the OMRON HEM-907XL automatic professional digital blood pressure monitor in mm Hg.
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
mm Hg | 122.54 (1.78) | 125.14 (1.71)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.292, Mixed Models Analysis

12. Primary Outcome: Diastolic Blood Pressure at 52 Weeks
Description: Measured by the OMRON HEM-907XL automatic professional digital blood pressure monitor in mm Hg.
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
mm Hg | 72.62 (1.22) | 74.06 (1.18)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.396, Mixed Models Analysis

13. Secondary Outcome: Subjective Functional Status at 25 Weeks
Description: Measured by the Physical Function subscale of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index; the subscale score range is 0-68; lower scores are better.
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale | 16.68 (1.44) | 18.30 (1.42)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.424, Mixed Models Analysis

14. Secondary Outcome: Quadriceps Strength at 25 Weeks
Description: Measured by the MicroFET2 hand-held dynamometer in terms of mean maximum pounds over two trials.
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: pounds
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
pounds | 43.21 (1.75) | 41.88 (1.71)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.586, Mixed Models Analysis

15. Secondary Outcome: Pain by the Pain Subscale of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index at 25 Weeks
Description: Measured by the Pain subscale of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index; the subscale score range is 0-20; lower scores are better.
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale | 4.25 (0.39) | 4.54 (0.38)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.596, Mixed Models Analysis

16. Secondary Outcome: Pain by the Bodily Pain Subscale of the Short Form-36v2 at 25 Weeks
Description: Measured by the Bodily Pain subscale of the Short Form-36v2; the subscale score range is 0-100; higher scores are better.
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale | 59.65 (2.32) | 58.13 (2.26)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.639, Mixed Models Analysis

17. Secondary Outcome: Fatigue at 25 Weeks
Description: Measured by the Brief Fatigue Inventory, which assesses fatigue severity; the scale score range is 0-10; lower scores are better.
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale | 2.49 (0.27) | 2.76 (0.25)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.466, Mixed Models Analysis

18. Secondary Outcome: Health-Related Quality of Life at 25 Weeks
Description: Measured by the Short Form-36v2 in terms of the following:
  Mental Component: this summary scale is composed of eight subscale scores primarily derived from the mental health, role functioning-emotional, and social functioning scores; the scale score range is 0-100; higher scores are better Physical Component: this summary scale is composed of eight subscale scores primarily derived from the physical functioning, role functioning-physical, and bodily pain scores; the scale score range is 0-100; higher scores are better
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale
  Short Form-36v2 Mental Component | 53.92 (1.11) | 52.30 (1.20)
  Short Form-36v2 Physical Component | 43.10 (0.97) | 43.07 (0.95)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.322, Mixed Models Analysis — p=0.322 for Short Form-36v2 Mental Component
Statistical Analysis 2: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.979, Mixed Models Analysis — p=0.979 for Short Form-36v2 Physical Component

19. Secondary Outcome: Self-Efficacy at 25 Weeks
Description: Measured by the Self-Efficacy Scale in terms of the following:
  Exercise Barriers Self-Efficacy subscale: the subscale score range is 0-100; higher scores are better Exercise Self-Efficacy subscale: the subscale score range is 0-100; higher scores are better
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale
  Exercise Barriers Self-Efficacy | 59.81 (2.77) | 58.37 (2.69)
  Exercise Self-Efficacy | 67.43 (3.44) | 60.20 (3.35)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.710, Mixed Models Analysis — p=0.710 for Exercise Barriers Self-Efficacy
Statistical Analysis 2: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.133, Mixed Models Analysis — p=0.133 for Exercise Self-Efficacy

20. Secondary Outcome: Arthritis Self-Efficacy at 25 Weeks
Description: Measured by the Arthritis Self-Efficacy Scale in terms of the following:
  Pain subscale: the subscale score range is 10-100; higher scores are better Function subscale: the subscale score range is 10-100; higher scores are better Other Symptoms subscale: the subscale score range is 10-100; higher scores are better
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale
  Arthritis Self Efficacy Pain | 75.58 (1.97) | 67.38 (2.13)
  Arthritis Self-Efficacy Function | 85.74 (1.79) | 85.90 (1.67)
  Arthritis Self-Efficacy Other Symptoms | 78.88 (1.99) | 77.66 (1.95)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.005, Mixed Models Analysis — p=0.005 for Arthritis Self Efficacy Pain
Statistical Analysis 2: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.948, Mixed Models Analysis — p=0.948 for Arthritis Self Efficacy Function
Statistical Analysis 3: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.663, Mixed Models Analysis — p=0.663 for Arthritis Self Efficacy Other Symptoms

21. Secondary Outcome: Outcome Expectancy at 25 Weeks
Description: Measured by the Perceived Therapeutic Efficacy Scale in terms of the following:
  Exercise and Arthritis: the scale score range is 0-100; higher scores are better Exercise and Hypertension: the scale score range is 0-100; higher scores are better
Time Frame: At the end of the 6-month intervention period (week 25)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale
  Perceived Therapeutic Efficacy Arthritis | 72.79 (2.41) | 59.67 (2.91)
  Perceived Therapeutic Efficacy Hypertension | 77.14 (2.48) | 69.62 (2.42)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.001, Mixed Models Analysis — p=0.001 for Perceived Therapeutic Efficacy of Exercise and Arthritis
Statistical Analysis 2: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.031, Mixed Models Analysis — p=0.031 for Perceived Therapeutic Efficacy of Exercise and Hypertension

22. Secondary Outcome: Subjective Functional Status at 52 Weeks
Description: as for outcome 13
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale | 17.02 (1.49) | 17.51 (1.44)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.816, Mixed Models Analysis

23. Secondary Outcome: Quadriceps Strength at 52 Weeks
Description: Measured by the MicroFET2 hand-held dynamometer in terms of mean maximum pounds over two trials.
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: pounds
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
pounds | 43.66 (1.77) | 43.33 (1.73)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.895, Mixed Models Analysis

24. Secondary Outcome: Pain by the Pain Subscale of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index at 52 Weeks
Description: as for outcome 15
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale | 4.09 (0.41) | 4.72 (0.39)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.260, Mixed Models Analysis

25. Secondary Outcome: Pain by the Bodily Pain Subscale of the Short Form-36v2 at 52 Weeks
Description: as for outcome 16
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale | 59.73 (2.36) | 59.70 (2.28)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.993, Mixed Models Analysis

26. Secondary Outcome: Fatigue at 52 Weeks
Description: as for outcome 17
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale | 2.97 (0.28) | 2.94 (0.25)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.947, Mixed Models Analysis

27. Secondary Outcome: Health-Related Quality of Life at 52 Weeks
Description: as for outcome 18
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale
  Short Form-36v2 Mental Component | 53.18 (1.12) | 51.81 (1.21)
  Short Form-36v2 Physical Component | 42.10 (1.18) | 42.47 (1.15)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.406, Mixed Models Analysis — p=0.406 for Short Form-36v2 Mental Component
Statistical Analysis 2: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.826, Mixed Models Analysis — p=0.826 for Short Form-36v2 Physical Component

28. Secondary Outcome: Self-Efficacy at 52 Weeks
Description: as for outcome 19
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale
  Exercise Barriers Self-Efficacy | 53.30 (2.83) | 53.05 (2.73)
  Exercise Self-Efficacy | 55.49 (3.56) | 51.00 (3.43)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.950, Mixed Models Analysis — p=0.950 for Exercise Barriers Self-Efficacy
Statistical Analysis 2: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.365, Mixed Models Analysis — p=0.365 for Exercise Self-Efficacy

29. Secondary Outcome: Arthritis Self-Efficacy at 52 Weeks
Description: as for outcome 20
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale
  Arthritis Self-Efficacy Pain | 73.15 (2.06) | 69.44 (2.19)
  Arthritis Self-Efficacy Function | 85.38 (1.82) | 87.75 (1.69)
  Arthritis Self-Efficacy Other Symptoms | 75.92 (2.03) | 75.23 (1.96)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.219, Mixed Models Analysis — p=0.219 for Arthritis Self Efficacy Pain
Statistical Analysis 2: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.340, Mixed Models Analysis — p=0.340 for Arthritis Self Efficacy Function
Statistical Analysis 3: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.806, Mixed Models Analysis — p=0.806 for Arthritis Self Efficacy Other Symptoms

30. Secondary Outcome: Outcome Expectancy at 52 Weeks
Description: as for outcome 21
Time Frame: 6 months after the intervention period ends (week 52)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STAR Intervention | Attention-Control
Number analyzed (Participants) | 91 | 91
units on a scale
  Perceived Therapeutic Efficacy Arthritis | 67.09 (2.83) | 55.86 (3.07)
  Perceived Therapeutic Efficacy Hypertension | 73.40 (2.53) | 67.93 (2.44)
Statistical Analysis 1: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.008, Mixed Models Analysis — p=0.008 for Perceived Therapeutic Efficacy of Exercise and Arthritis
Statistical Analysis 2: Comparison: STAR Intervention vs Attention-Control; Test type: Superiority; p = 0.120, t-test, 1 sided — p=0.120 for Perceived Therapeutic Efficacy of Exercise and Hypertension

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | STAR Intervention | Attention-Control
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/91
Other Adverse Events (participants affected / at risk) | 0/91 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No